CLINICAL TRIAL: NCT04980924
Title: Pulmonary Embolism Registry
Brief Title: Epidemiology and Clinical Course of Pulmonary Embolism During and After Hospitalisation
Acronym: REMATEV
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 21cardio01
Record Dates: First submitted 2021-07-21; First posted 2021-07-28 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pulmonary Embolism without reccurence or complication: Pulmonary Embolism without reccurence or complication
  Interventions: Other: no intervention
- Pulmonary Embolism with reccurence or complication: Pulmonary Embolism with reccurence or complication, in particular occurrence of pulmonary hypertension.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
This survey will allow to identify PE prognostic, but also long-term complications, i.e. recurrence rate, on-treatment bleedings, deep-vein thrombosis sequella, pulmonary hypertension rate, and chronic pulmonary disease rate without PH. This database should help us identify risk-factors for each event.

ELIGIBILITY:
Inclusion Criteria:

* All pulmonary embolisms hospitalised in Nice hospital.
* acceptation to enter in the cohorte survey

Exclusion Criteria:

-

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All pulmonary embolisms hospitalised in our department
Sampling Method: Non-Probability Sample
Enrollment: 547 (Actual)
Dates: Start 1992-01-01 (Actual); Primary Completion 1997-12-31 (Actual); Study Completion 1997-12-31 (Actual)

PRIMARY OUTCOMES:
Reccurence | 10 years
  number of patient with Documented symptomatic pulmonary embolism reccurence

SECONDARY OUTCOMES:
Pulmonary hypertension | 10 years
  number of patients with Confirmed pulmonary hypertension after pulmonary embolism
Chronic pulmonary disease without hypertension | 10 years
  number of patients with dyspnea but without pulmonary hypertension, Documented non-reperfused pulmonary areas

CONTACTS AND LOCATIONS:
Locations (1):
- Nice University Hospital, Nice, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ferrari E, Fourrier E, Asarisi F, Heme N, Redjimi N, Berkane N, Labbaoui M, Breittmayer JP, Bun SS, Moceri P, Squara F. Is pulmonary embolism recurrence linked with the severity of the first event? A French retrospective cohort study. BMJ Open. 2021 Sep 29;11(9):e050910. doi: 10.1136/bmjopen-2021-050910. PMID 34588255